CLINICAL TRIAL: NCT00861211
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Assess The Safety and Efficacy of Two Weeks of Oral Senicapoc Administration on Allergen Challenge in Atopic Asthmatic Subjects
Brief Title: Safety and Efficacy Study of Oral Senicapoc on Allergen Challenge in Atopic Asthmatic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Icagen (Industry)
Responsible Party: Seth V. Hetherington, M.D. Sr. VP Clinical and Regulatory Affairs, Icagen, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ICA-17043-17
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Atopic Asthma
Keywords: asthma; inflammation; bronchoconstriction; allergen challenge; KCa3.1
MeSH Terms: conditions — Asthma; Inflammation | interventions — senicapoc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active treatment arm (Experimental)
  Interventions: Drug: senicapoc
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: senicapoc — Loading Dose: 80 mg twice daily x 3 days followed by Maintenance Dose: 40 mg daily x 11 days
  Other Names: ICA-17043
  Arms: Active treatment arm
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether senicapoc can decrease changes in FEV1 following allergen challenge in atopic allergic subjects.

DETAILED DESCRIPTION:
Based on the unmet medical need for new agents in the treatment of asthma and the role of KCa3.1 in the function of several different cell types involved in the inflammatory response, and the effects seen in an animal model of allergic asthma, it is reasonable to explore the utility of senicapoc, a KCa3.1 blocker, as a novel treatment of asthma. This study will test the ability of senicapoc to alleviate bronchospasm induced by an allergen challenge in patients with allergic asthma. It is analogous to the study performed in animals in which senicapoc demonstrated the ability to reduce airway resistance and hyper-responsiveness induced by airway challenge with antigen and carbachol, respectively. This study is also the first to test the ability of senicapoc to reduce airway inflammation, which is the key pathophysiologic process in asthma. In summary, with a demonstrated safety profile across a wide range of doses in humans and efficacy in an animal model of allergic bronchospasm and hyper-responsiveness, the initiation of exploratory studies of senicapoc for treatment of asthma is justified.

ELIGIBILITY:
Inclusion Criteria:

* History of asthma (as defined by the Global Initiative in Asthma definition or having been previously treated for asthma);
* Baseline (pre-bronchodilator) forced expiratory volume at one second (FEV1) ≥70% of predicted;
* Clinically acceptable medical history, physical examination, 12 lead ECG, vital signs, and clinical laboratory tests );
* Positive response on screening to skin prick test to either house dust mite, cat hair, or grass pollen;
* A positive inhaled methacholine challenge with a PC20 ≤ 8 mg/mL (within 6 months prior to Screening Visit 1);
* Screening allergen challenge demonstrates that the subject experiences both an early and late asthmatic response. The early asthmatic response must include a fall in FEV1 of equal to or more than 20% from the post saline value, on at least one occasion, between 5 and 30 minutes after the final concentration of allergen. The late asthmatic response must include a fall in FEV1 of equal to or more than 15% from the post saline value, on at least three occasions, two of which must be consecutive, between 4 and 10 hours after the final concentration of allergen;
* Non-smoker (refrained from any tobacco usage or any products containing nicotine for 6 months prior to Screening Visit 1);
* Able and willing to give written informed consent to participate in the study.

Exclusion Criteria:

* Any subject who has experienced any allergic reaction to a drug that suggests an increased potential for a hypersensitivity to senicapoc (e.g. clotrimazole);
* Previous ingestion of senicapoc (ICA-17043) prior to Screening Visit 1;
* Any condition that might interfere with the absorption, distribution, metabolism, and/or excretion of drugs;
* Respiratory tract infection or asthma exacerbation within 4 weeks of the first Screening Visit or within the period between Screening Visit 1 and Day 1 unless study physician believes lung function was unaffected (no greater than 10% decrease in baseline FEV1) by such event;
* Considering or scheduled to undergo any surgical procedure during the duration of the study;
* History of alcohol and/or drug abuse within 2 years prior to Screening Visit 1;
* Donation of blood (>450 mL) or significant loss of blood within 56 days prior to Screening Visit 1;
* Received any commercially licensed investigational product within 30 days prior to Screening Visit 1 or received any unlicensed investigational product within 90 days prior to Screening Visit 1;
* History of chronic hepatitis B or C, a positive test for hepatitis B surface antigen, hepatitis C antibody, a history of HIV infection, or demonstration of HIV antibodies;
* A positive qualitative urine drug test, a positive urine or breath alcohol test, or a positive urine cotinine or CO breath test at the first Screening visit or on Day 1;
* Use of oral or inhaled or intranasal corticosteroid, long acting beta agonists (e.g., salmeterol or formoterol), leukotriene receptor antagonists (e.g., zafirlukast or montelukast), theophylline, nedocromil sodium, cromolyn sodium, zileuton , or anti-cholinergic agents within the 28 days prior to the first Screening visit;
* Use of oral antihistamines within 1 week prior to the first Screening visit;
* Symptomatic with hay fever during any of the Screening Visits or Day 1;
* A >10 pack year cigarette history.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Decrease in FEV1 between 4-10 hours (Late Asthmatic Response) after allergen challenge and will compare the active (40 mg QD) vs. placebo treatment groups with respect to change in response to allergen challenge. | after 2 weeks of treatment with study medication

SECONDARY OUTCOMES:
Early allergen response to allergen challenge, measure of airway hyperreactivity to methacholine challenge, pulmonary function tests (FEV1 and FVC), fraction of exhaled NO, cell differentials and cytokine measurements from induced sputum samples. | after 2 weeks of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Tak H Lee, FRCP, Principal Investigator — Guy's Drug Research Unit, Quintiles Limited
Locations (2):
- United Kingdom (2):
  - Guy's Drug Research Unit, London, UK
  - Medicines Evaluation Unit, Manchester, UK